CLINICAL TRIAL: NCT03813641
Title: Phase Ⅱ Clinical Study of RALOX or CAPOX Combined With Bevacizumab in the First-line Treatment of Advanced Colorectal Cancer
Brief Title: RALOX or CAPOX + Bevacizumab in the First-line Treatment of Advanced CRC(ROCB Study)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Principal Investigator, Ruilian Xu, Phase Ⅱ Clinical Study of RALOX or CAPOX Combined With Bevacizumab in the First-line Treatment of Advanced Colorectal Cancer, Shenzhen People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Shenzhen CRC-002
Record Dates: First submitted 2019-01-20; First posted 2019-01-23 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Colorectal Cancer
Keywords: Raltitrexed; First-line therapy; Bevacizumab; Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — raltitrexed; Capecitabine

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RALOX + bevacizumab (Experimental): Oxaliplatin 130mg/m2, i.v.gtt 2h, d1 Raltitrexed 3mg/m2, i.v.gtt 15min ,d1 Bevacizumab 7.5mg/kg, i.v.gtt, d1 The above schemes are repeated every three weeks. After 8 cycles, such as CR, PR or SD, the regimen is changed to raltitrexed (3mg/m2, intravenous drip for 15 minutes, d1)+bevacizumab (7.5mg/kg, intravenous drip, d1). The regimen is repeated every 3 weeks until the disease progresses.
  Interventions: Drug: Raltitrexed
- CAPOX + bevacizumab (Active Comparator): Oxaliplatin 130mg/m2, i.v.gtt 2h, d1 Capecitabine 1000mg/m2, po. ,d1 Bevacizumab 7.5mg/kg, i.v.gtt, d1 The above schemes are repeated every three weeks. After 8 cycles, such as CR, PR or SD, the regimen is changed to Capecitabine (1000mg/m2 po. d1-14)+bevacizumab (7.5mg/kg, intravenous drip, d1). The regimen is repeated every 3 weeks until the disease progresses.
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Raltitrexed — Experimental: Oxaliplatin + Raltitrexed + Bevacizumab The above schemes are repeated every three weeks. After 8 cycles, such as CR, PR or SD, the regimen is changed to Raltitrexed (3mg/m2, intravenous drip for 15 minutes, d1)+bevacizumab (7.5mg/kg, intravenous drip, d1). The regimen is repeated every 3 weeks until the disease progresses.
  Other Names: Tomudex
  Arms: RALOX + bevacizumab
Drug: Capecitabine — Other: Oxaliplatin + Capecitabine + Bevacizumab The above schemes are repeated every three weeks. After 8 cycles, such as CR, PR or SD, the regimen is changed to Capecitabine (1000mg/m2 po. d1-14)+bevacizumab (7.5mg/kg, intravenous drip, d1). The regimen is repeated every 3 weeks until the disease progresses.
  Other Names: Xeloda
  Arms: CAPOX + bevacizumab

SUMMARY:
Raltitrexed is an inhibitor of thymidylate synthase.As a folate antimetabolite drug, raltitrexed has been used in treatment of colorectal cancer(CRC) since 1998, and also used in malignant mesothelioma.Several phase III studies performed in patients with advanced CRC showed that it is as effective as 5-fluorouracil(5-FU) /leucovorin(LV) with regard to response rates and survival. The combination of raltitrexed with oxaliplatin shows response rates of 41%-54% and median survivals of 14.6-14.8 months, which are comparable to those achieved with 5-FU/LV combination with oxaliplatin. This study discussed the efficacy and safety of raltitrexed-oxaliplatin(RALOX) combined with bevacizumab or capecitabine-oxaliplatin(CAPOX) combined with bevacizumab in first-line treatment of patients with advanced colorectal cancer who could not undergo radical surgery. The main endpoint will be progression free survival (PFS). The secondary endpoints will be overall survival, objective response rate and disease control rate (OS,ORR and DCR).It is expected that raltitrexed may be one of options for the treatment of advanced CRC in the first-line setting.

DETAILED DESCRIPTION:
According to the inclusion and exclusion criteria, the patients will be randomly divided into two groups: the experimental group (group A) will be administered with raltitrexed 3mg/m2 intravenously combined with oxaliplatin and bevacizumab, repeated every 21 days. The control group (group B) will be administered with orally capecitabine (1000mg/m2, d 1-14) combined with oxaliplatin and bevacizumab, repeated every 21 days. After 8 cycles of treatments, if evaluated as complete response(CR),partial response(PR) or stable disease(SD), CRC patients will go into maintenance therapy wtih raltitrexed combined with bevacizumab in group A or capecitabine combined with bevacizumab in group B respectively, ended in disease progression(PD) , symptoms deterioration, unacceptable toxicity, death or withdrawal of consent (whichever occurs first). The radiological efficacy will be evaluated every 6 weeks (2 treatment cycles) and non-PD (PD criteria referring to RECIST 1.1 criteria) patients will continue to be treated until the cancer progression or the patient's intolerable toxicity or death. Toxic side effects and quality of life will be assessed at the same time.

Follow up participants and analyse primary endpoint (PFS) and secondary endpoints (OS,ORR and DCR).The causes of confirmed missing data in the trial should be recorded in detail to determine the mechanism of missing data and choose the suitable missing data handling methods.

ELIGIBILITY:
Inclusion Criteria:

* Age 18~75 years;
* Patients are diagnosed by histopathological and/or cytological examination as local advanced or metastatic colorectal cancer who are unable to undergo radical surgery with no symptom of the primary lesions；
* There are one or more measurable lesions, the longest diameter of which is at least 10 mm by spiral CT scanning (RECIST standard, version 1.1)
* ECOG performance status (ECOG PS) 0~1;
* Life expectancy not less than 3 month
* Blood routine, liver and kidney function reached the following criteria within 14 days before screening:

Absolute neutrophil count (> 1.5x109/L); hemoglobin (> 9.0 g/dl); platelet count (> 100 x109/L); total bilirubin (< 1.5 times the normal upper limit (ULN); alanine aminotransferase and glutamic oxaloacetate aminotransferase (< 2.5 x ULN) in patients with liver metastasis (< 5 x ULN); alkaline phosphatase （< 3 x ULN（ in patients with liver metastasis < 5 x ULN)）; serum creatinine （< 1.5 x ULN）;

* Adequate blood coagulation function [International Normalized Ratio (INR) ≤1.5 and Partial Thromboplastin Time (PTT) or activated PTT (aPTT) ≤1.5 x upper limit of normal (ULN)). Participants on full-dose anticoagulation must be in a stable phase of anticoagulant therapy and if taking oral anticoagulation, participants must have an INR ≤3 without clinically significant active bleeding or a high risk of bleeding.
* Agree to provide histological specimens from previous operations for biomarker assessment and specimens remain。
* Signed informed consent to be provided

Exclusion Criteria:

* Previous treatment with Raltitrexed；
* With a large amount of pleural effusions or ascites requiring puncture drainage；
* Active clinical severe infections include hepatitis；
* One of the following complications: 1) Gastrointestinal obstruction (including paralytic ileus) or gastrointestinal bleeding 2) Symptomatic cardiac disease (including unstable angina, myocardial infarction, and heart failure) 3) Pulmonary fibrosis or interstitial pneumonia 4) Uncontrolled diabetes mellitus 5) Uncontrolled diarrhea (that affects daily activities although adequate therapy )
* Symptomatic brain or meningeal metastasis (unless the patient has been treated for > 6 months, the imaging results are negative in the 4 weeks before entering the study, and the clinical symptoms associated with the tumor are stable at the time of entering the study);
* Undergoing kidney dialysis；
* History of other malignant tumors within 5 years, except for cured cervical carcinoma in situ or basal cell carcinoma of the skin;
* Drug abuse and medical, psychological or social conditions may interfere with patients' participation in the study or have an impact on the evaluation of the study results；
* Pregnant or lactating females, and males and females reluctant to use contraception
* History of concurrent gastrointestinal perforation or gastrointestinal perforation within 1 year prior to enrollment
* Pulmonary hemorrhage/hemoptysis ≥ Grade 2 (identified as bright red blood of not less 2.5mL) within 1 month before enrollment.
* History of thoracotomy,laparotomy, or intestinal resection within 28 days prior to enrollment;
* Unhealed wound (other than suture wounds due to implantation of a central venous port), traumatic fracture, or gastrointestinal ulcer
* Current cerebrovascular disease or thromboembolism or either within 1 year before enrollment
* Current anticoagulation therapy or requiring anticoagulation agents (> 325 mg/day of aspirin)
* Bleeding diathesis, coagulopathy, or coagulation factor abnormality (INR ≥1.5 within 14 days before enrollment)
* Uncontrolled hypertension
* Urine dipstick for proteinuria >+2
* Researchers think those should be excluded

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-01-28 (Actual); Primary Completion 2021-02-28 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) Time | The follow-up period ranges from the first patient recruited to the last patient within 6 months after admission, up to 2 years.
  PFS is defined as the time from the date of randomization until the date of objectively determined progressive disease (PD) [according to Response Evaluation Criteria in Solid Tumors (RECIST) version (v). 1.1] or death due to any cause, whichever will be first. PD is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 millimeters (mm). Participants who died without a reported prior progression will be considered to have progressed on the day of their death. Participants who do not progress or be lost to follow-up will be censored at the day of their last radiographic tumor assessment.

SECONDARY OUTCOMES:
Overall Survival (OS) | The follow-up period ranges from the first patient recruited to the last patient within 6 months after admission,up to 2 years.
  OS is defined as the time in months from the date of randomization to the date of death from any cause. For participants not known to have died as of the cut-off date, OS will be censored at the last known date alive.
Percentage of Participants Achieving an Objective Response (Objective Response Rate) | The follow-up period ranges from the first patient recruited to the last patient within 3 months after admission.
  The objective response rate is equal to the proportion of participants achieving a best overall response of partial response or complete response (PR + CR). Response is defined using RECIST, v. 1.1 criteria. CR is defined as the disappearance of all target and non-target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm and normalization of tumor marker level of non-target lesions; PR is defined as having at least a 30% decrease in sum of longest diameter of target lesions taking as reference the baseline sum diameter.
Percentage of Participants Achieving a Stable Disease (SD) or a confirmed CR or PR (Disease Control Rate) | The follow-up period ranges from the first patient recruited to the last patient within 3 months after admission.
  Participants achieved disease control if they have a best overall response of CR, PR or SD. According to RECIST v1.1, CR is the disappearance of all non-nodal target lesions, with the short axes of any target lymph node reduced to <10 mm, the disappearance of all non-target lesions, and the normalization of tumor marker levels (if tumor markers were initially above the ULN); PR was defined as at least a 30% decrease in the sum of the diameters of target lesions (including the short axes of any target lymph node), taking as reference the baseline sum diameter. SD is neither sufficient shrinkage to qualify as PR nor sufficient increase to qualify as PD, taking as reference the smallest sum diameter since treatment started.

CONTACTS AND LOCATIONS:
Overall Officials: Ruilian Xu, MD, Principal Investigator — Shen Zhen People's Hospital
Locations (1):
- Shenzhen People's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kindler HL, Shulman KL. Metastatic colorectal cancer. Curr Treat Options Oncol. 2001 Dec;2(6):459-71. doi: 10.1007/s11864-001-0068-7. PMID 12057092
- [Background] Meta-analysis Group In Cancer; Piedbois P, Rougier P, Buyse M, Pignon J, Ryan L, Hansen R, Zee B, Weinerman B, Pater J, Leichman C, Macdonald J, Benedetti J, Lokich J, Fryer J, Brufman G, Isacson R, Laplanche A, Levy E. Efficacy of intravenous continuous infusion of fluorouracil compared with bolus administration in advanced colorectal cancer. J Clin Oncol. 1998 Jan;16(1):301-8. doi: 10.1200/JCO.1998.16.1.301. PMID 9440757
- [Background] Modulation of fluorouracil by leucovorin in patients with advanced colorectal cancer: evidence in terms of response rate. Advanced Colorectal Cancer Meta-Analysis Project. J Clin Oncol. 1992 Jun;10(6):896-903. doi: 10.1200/JCO.1992.10.6.896. PMID 1534121
- [Background] Meta-Analysis Group In Cancer; Levy E, Piedbois P, Buyse M, Pignon JP, Rougier P, Ryan L, Hansen R, Zee B, Weinerman B, Pater J, Leichman C, Macdonald J, Benedetti J, Lokich J, Fryer J, Brufman G, Isacson R, Laplanche A, Quinaux E, Thirion P. Toxicity of fluorouracil in patients with advanced colorectal cancer: effect of administration schedule and prognostic factors. J Clin Oncol. 1998 Nov;16(11):3537-41. doi: 10.1200/JCO.1998.16.11.3537. PMID 9817272
- [Background] Becker K, Erckenbrecht JF, Haussinger D, Frieling T. Cardiotoxicity of the antiproliferative compound fluorouracil. Drugs. 1999 Apr;57(4):475-84. doi: 10.2165/00003495-199957040-00003. PMID 10235688
- [Background] Wacker A, Lersch C, Scherpinski U, Reindl L, Seyfarth M. High incidence of angina pectoris in patients treated with 5-fluorouracil. A planned surveillance study with 102 patients. Oncology. 2003;65(2):108-12. doi: 10.1159/000072334. PMID 12931015
- [Background] Rougier P, Van Cutsem E, Bajetta E, Niederle N, Possinger K, Labianca R, Navarro M, Morant R, Bleiberg H, Wils J, Awad L, Herait P, Jacques C. Randomised trial of irinotecan versus fluorouracil by continuous infusion after fluorouracil failure in patients with metastatic colorectal cancer. Lancet. 1998 Oct 31;352(9138):1407-12. doi: 10.1016/S0140-6736(98)03085-2. PMID 9807986
- [Background] Cunningham D, Pyrhonen S, James RD, Punt CJ, Hickish TF, Heikkila R, Johannesen TB, Starkhammar H, Topham CA, Awad L, Jacques C, Herait P. Randomised trial of irinotecan plus supportive care versus supportive care alone after fluorouracil failure for patients with metastatic colorectal cancer. Lancet. 1998 Oct 31;352(9138):1413-8. doi: 10.1016/S0140-6736(98)02309-5. PMID 9807987
- [Background] Seymour MT, Maughan TS, Ledermann JA, Topham C, James R, Gwyther SJ, Smith DB, Shepherd S, Maraveyas A, Ferry DR, Meade AM, Thompson L, Griffiths GO, Parmar MK, Stephens RJ; FOCUS Trial Investigators; National Cancer Research Institute Colorectal Clinical Studies Group. Different strategies of sequential and combination chemotherapy for patients with poor prognosis advanced colorectal cancer (MRC FOCUS): a randomised controlled trial. Lancet. 2007 Jul 14;370(9582):143-152. doi: 10.1016/S0140-6736(07)61087-3. PMID 17630037
- [Background] Graeven U, Arnold D, Reinacher-Schick A, Heuer T, Nusch A, Porschen R, Schmiegel W. A randomised phase II study of irinotecan in combination with 5-FU/FA compared with irinotecan alone as second-line treatment of patients with metastatic colorectal carcinoma. Onkologie. 2007 Apr;30(4):169-74. doi: 10.1159/000099636. Epub 2007 Mar 23. PMID 17396039
- [Background] Leonard P, Seymour MT, James R, Hochhauser D, Ledermann JA. Phase II study of irinotecan with bolus and high dose infusional 5-FU and folinic acid (modified de Gramont) for first or second line treatment of advanced or metastatic colorectal cancer. Br J Cancer. 2002 Nov 18;87(11):1216-20. doi: 10.1038/sj.bjc.6600641. PMID 12439708
- [Background] Rougier P, Lepille D, Bennouna J, Marre A, Ducreux M, Mignot L, Hua A, Mery-Mignard D. Antitumour activity of three second-line treatment combinations in patients with metastatic colorectal cancer after optimal 5-FU regimen failure: a randomised, multicentre phase II study. Ann Oncol. 2002 Oct;13(10):1558-67. doi: 10.1093/annonc/mdf259. PMID 12377643
- [Background] Peeters M, Price TJ, Cervantes A, Sobrero AF, Ducreux M, Hotko Y, Andre T, Chan E, Lordick F, Punt CJ, Strickland AH, Wilson G, Ciuleanu TE, Roman L, Van Cutsem E, Tzekova V, Collins S, Oliner KS, Rong A, Gansert J. Randomized phase III study of panitumumab with fluorouracil, leucovorin, and irinotecan (FOLFIRI) compared with FOLFIRI alone as second-line treatment in patients with metastatic colorectal cancer. J Clin Oncol. 2010 Nov 1;28(31):4706-13. doi: 10.1200/JCO.2009.27.6055. Epub 2010 Oct 4. PMID 20921462
- [Background] Fuchs CS, Marshall J, Mitchell E, Wierzbicki R, Ganju V, Jeffery M, Schulz J, Richards D, Soufi-Mahjoubi R, Wang B, Barrueco J. Randomized, controlled trial of irinotecan plus infusional, bolus, or oral fluoropyrimidines in first-line treatment of metastatic colorectal cancer: results from the BICC-C Study. J Clin Oncol. 2007 Oct 20;25(30):4779-86. doi: 10.1200/JCO.2007.11.3357. PMID 17947725
- [Background] Tournigand C, Andre T, Achille E, Lledo G, Flesh M, Mery-Mignard D, Quinaux E, Couteau C, Buyse M, Ganem G, Landi B, Colin P, Louvet C, de Gramont A. FOLFIRI followed by FOLFOX6 or the reverse sequence in advanced colorectal cancer: a randomized GERCOR study. J Clin Oncol. 2004 Jan 15;22(2):229-37. doi: 10.1200/JCO.2004.05.113. Epub 2003 Dec 2. PMID 14657227
- [Background] Jarmula A. Antifolate inhibitors of thymidylate synthase as anticancer drugs. Mini Rev Med Chem. 2010 Nov;10(13):1211-22. doi: 10.2174/13895575110091211. PMID 20854257
- [Background] Wilson KS, Malfair Taylor SC. Raltitrexed: optimism and reality. Expert Opin Drug Metab Toxicol. 2009 Nov;5(11):1447-54. doi: 10.1517/17425250903307455. PMID 19863453
- [Background] Cunningham D. Mature results from three large controlled studies with raltitrexed ('Tomudex'). Br J Cancer. 1998;77 Suppl 2(Suppl 2):15-21. doi: 10.1038/bjc.1998.421. PMID 9579851
- [Background] Cocconi G, Cunningham D, Van Cutsem E, Francois E, Gustavsson B, van Hazel G, Kerr D, Possinger K, Hietschold SM. Open, randomized, multicenter trial of raltitrexed versus fluorouracil plus high-dose leucovorin in patients with advanced colorectal cancer. Tomudex Colorectal Cancer Study Group. J Clin Oncol. 1998 Sep;16(9):2943-52. doi: 10.1200/JCO.1998.16.9.2943. PMID 9738562
- [Background] Feliu J, Mel JR, Camps C, Escudero P, Aparicio J, Menendez D, Garcia Giron C, Rodriguez MR, Sanchez JJ, Gonzalez Baron M; Oncopaz Cooperative Group Associated Hospitals. Raltitrexed in the treatment of elderly patients with advanced colorectal cancer: an active and low toxicity regimen. Eur J Cancer. 2002 Jun;38(9):1204-11. doi: 10.1016/s0959-8049(02)00005-9. PMID 12044507
- [Background] Cascinu S, Graziano F, Ferrau F, Catalano V, Massacesi C, Santini D, Silva RR, Barni S, Zaniboni A, Battelli N, Siena S, Giordani P, Mari D, Baldelli AM, Antognoli S, Maisano R, Priolo D, Pessi MA, Tonini G, Rota S, Labianca R. Raltitrexed plus oxaliplatin (TOMOX) as first-line chemotherapy for metastatic colorectal cancer. A phase II study of the Italian Group for the Study of Gastrointestinal Tract Carcinomas (GISCAD). Ann Oncol. 2002 May;13(5):716-20. doi: 10.1093/annonc/mdf091. PMID 12075739
- [Background] Cortinovis D, Bajetta E, Di Bartolomeo M, Dognini G, Beretta E, Ferrario E, Ricotta R, Buzzoni R. Raltitrexed plus oxaliplatin in the treatment of metastatic colorectal cancer. Tumori. 2004 Mar-Apr;90(2):186-91. doi: 10.1177/030089160409000205. PMID 15237580
- [Background] Laudani A, Gebbia V, Leonardi V, Savio G, Borsellino N, Cusimano MP, Calabria C, Stefano R, Agostara B. Activity and toxicity of oxaliplatin plus raltitrexed in 5-fluorouracil refractory metastatic colorectal adeno-carcinoma. Anticancer Res. 2004 Mar-Apr;24(2C):1139-42. PMID 15154638
- [Background] Santini D, Massacesi C, D'Angelillo RM, Marcucci F, Campisi C, Vincenzi B, Pilone A, Bianco V, Bonsignori M, Tonini G. Raltitrexed plus weekly oxaliplatin as first-line chemotherapy in metastatic colorectal cancer: a multicenter non-randomized phase ii study. Med Oncol. 2004;21(1):59-66. doi: 10.1385/MO:21:1:59. PMID 15034215
- [Background] Martoni A, Mini E, Pinto C, Gentile AL, Nobili S, Dentico P, Marino A, Scicolone S, Angelelli B, Mazzei T. Oxaliplatin plus raltitrexed in the treatment of patients with advanced colorectal cancer: a phase II study. Anticancer Res. 2003 Jan-Feb;23(1B):687-91. PMID 12680168
- [Background] Neri B, Doni L, Fulignati C, Perfetto F, Turrini M, Andreoli F, Pantalone D, Pernice LM, Taruffi F, Martini V, Poma A, Valeri A, Bacci G, Sancez L, Moretti R. Raltitrexed plus oxaliplatin as first-line chemotherapy in metastatic colorectal carcinoma: a multicentric phase II trial. Anticancer Drugs. 2002 Aug;13(7):719-24. doi: 10.1097/00001813-200208000-00006. PMID 12187328
- [Background] Scheithauer W, Kornek GV, Schuell B, Ulrich-Pur H, Penz M, Raderer M, Lang F, Schneeweiss B, Lenauer A, Depisch D. Second-line treatment with oxaliplatin + raltitrexed in patients with advanced colorectal cancer failing fluoropyrimidine/leucovorin-based chemotherapy. Ann Oncol. 2001 May;12(5):709-14. doi: 10.1023/a:1011194712661. PMID 11432632
- [Background] Gravalos C, Salut A, Garcia-Giron C, Garcia-Carbonero R, Leon AI, Sevilla I, Maurel J, Esteban B, Garcia-Rico E, Murias A, Cortes-Funes H. A randomized phase II study to compare oxaliplatin plus 5-fluorouracil and leucovorin (FOLFOX4) versus oxaliplatin plus raltitrexed (TOMOX) as first-line chemotherapy for advanced colorectal cancer. Clin Transl Oncol. 2012 Aug;14(8):606-12. doi: 10.1007/s12094-012-0843-x. Epub 2012 Jul 19. PMID 22855138
- [Background] Feliu J, Castanon C, Salud A, Mel JR, Escudero P, Pelegrin A, Lopez-Gomez L, Ruiz M, Gonzalez E, Juarez F, Lizon J, Castro J, Gonzalez-Baron M; Oncopaz Cooperative Group, Spain. Phase II randomised trial of raltitrexed-oxaliplatin vs raltitrexed-irinotecan as first-line treatment in advanced colorectal cancer. Br J Cancer. 2005 Nov 28;93(11):1230-5. doi: 10.1038/sj.bjc.6602860. PMID 16265344
- [Background] Cheng K, Chen Y, Li LH, Liu JY. Raltitrexed combined with bevacizumab in heavily pretreated metastatic colorectal cancer. J Cancer Res Ther. 2013 Oct-Dec;9(4):727-9. doi: 10.4103/0973-1482.126470. PMID 24518728
- [Background] Ito Y, Osaki Y, Tokudome N, Sugihara T, Takahashi S, Iwase T, Hatake K. Efficacy of S-1 in heavily pretreated patients with metastatic breast cancer: cross-resistance to capecitabine. Breast Cancer. 2009;16(2):126-31. doi: 10.1007/s12282-008-0073-9. Epub 2008 Sep 20. PMID 18807123
- [Background] Hoff PM, Pazdur R, Lassere Y, Carter S, Samid D, Polito D, Abbruzzese JL. Phase II study of capecitabine in patients with fluorouracil-resistant metastatic colorectal carcinoma. J Clin Oncol. 2004 Jun 1;22(11):2078-83. doi: 10.1200/JCO.2004.05.072. PMID 15169794
- [Background] Sato A, Kurihara M, Horikoshi N, Aiba K, Kikkawa N, Shirouzu K, Mitachi Y, Sakata Y, Wakui A. Phase II study of raltitrexed (Tomudex) in chemotherapy-pretreated patients with advanced colorectal cancer. Tomudex Cooperative Study Group. Anticancer Drugs. 1999 Sep;10(8):741-8. doi: 10.1097/00001813-199909000-00008. PMID 10573207
- [Background] Douillard JY, Siena S, Cassidy J, Tabernero J, Burkes R, Barugel M, Humblet Y, Bodoky G, Cunningham D, Jassem J, Rivera F, Kocakova I, Ruff P, Blasinska-Morawiec M, Smakal M, Canon JL, Rother M, Oliner KS, Tian Y, Xu F, Sidhu R. Final results from PRIME: randomized phase III study of panitumumab with FOLFOX4 for first-line treatment of metastatic colorectal cancer. Ann Oncol. 2014 Jul;25(7):1346-1355. doi: 10.1093/annonc/mdu141. Epub 2014 Apr 8. PMID 24718886